CLINICAL TRIAL: NCT00934674
Title: A Single Dose Bioequivalence Study Comparing the Commercial Tablet Formulation to the Clinical Tablet of Bosutinib in Healthy Subjects
Brief Title: Study Comparing Two Different Tablet Formulations Of Bosutinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3160A4-1115
Record Dates: First submitted 2009-07-02; First posted 2009-07-08 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: Healthy Subjects
MeSH Terms: interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Commercial Tablet manufactured by Excella
  Interventions: Drug: SKI-606 (Bosutinib)
- 2 (Experimental): Clinical Tablet manufactured by Wyeth Montreal
  Interventions: Drug: SKI-606 (Bosutinib)

INTERVENTIONS:
Drug: SKI-606 (Bosutinib) — Arm 1 - Commercial Tablet manufactured by Excella
  Arm 2 - Clinical Tablet manufactured by Wyeth Montreal
  Other Names: Bosutinib

SUMMARY:
This study is comparing 2 formulations of bosutinib in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of non-childbearing potential, age 18 to 50 years.

Exclusion Criteria:

* Any significant cardiovascular, renal, hepatic, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics as measured by Cmax, AUC, tmax, and t1/2 | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Tacoma, Washington, United States